CLINICAL TRIAL: NCT00779246
Title: Cost-Effectiveness of Chlorhexidine Bathing vs. Active Surveillance Cultures to Prevent Acquisition of Methicillin-resistant Staphylococcus Aureus and Other Hospital-Acquired Infections: A Pilot Study
Brief Title: Cost-Effectiveness Study Comparing Chlorhexidine Bathing With Active Surveillance Cultures to Prevent Methicillin-resistant Staphylococcus Aureus & Other Hospital Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: Sage Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 28116
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2012-03-21 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Staphylococcal Infections
Keywords: Methicillin resistance; Infection control; Staphylococcus aureus; Cross infection; Epidemiology; Chlorhexidine
MeSH Terms: conditions — Staphylococcal Infections; Cross Infection | interventions — chlorhexidine gluconate; Quarantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Active surveillance cultures (ASC) (via nasal swabs) will be performed for all patients admitted to the medical intensive care unit (ICU) during the designated study period. All patients will be placed in contact isolation until nasal swabs return negative; otherwise will remain in isolation.
  Interventions: Other: Nasal swabs for MRSA culture; Other: Contact isolation
- 2 (Active Comparator): Chlorhexidine gluconate (CHG) cloths will be used to bathe patients daily instead of standard soap and water. Active surveillance cultures (ASC) will also be used in this arm, but results will be blinded and not used to determine whether patients should be in contact isolation.
  Interventions: Other: Nasal swabs for MRSA culture; Drug: Chlorhexidine gluconate

INTERVENTIONS:
Other: Nasal swabs for MRSA culture — Patients will have nasal swabs performed upon ICU admission, upon discharge, and every 2 weeks while they remain in the ICU.
Drug: Chlorhexidine gluconate — CHG-impregnated cloths (2%) will be used to bathe patients at least daily during the duration of their medical ICU stay. Surveillance cultures will be obtained on admission, discharge and every 2 weeks while in the ICU, but results will be blinded until conclusion of the study.
  Other Names: Sage 2% Chlorhexidine gluconate cloth
  Arms: 2
Other: Contact isolation — All patients will be placed in contact isolation until the results of their active surveillance cultures are negative; if positive, they will remain in isolation.
  Arms: 1

SUMMARY:
This pilot study in our medical intensive care unit will evaluate the clinical and cost-effectiveness of an active surveillance program for methicillin-resistant Staphylococcus aureus (MRSA), compared to routine daily bathing with chlorhexidine gluconate (CHG)-impregnated cloths. Outcomes include rate of MRSA acquisition, and of other hospital-acquired infections (e.g., catheter-associated bloodstream infections).

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the medical intensive care unit (ICU) are eligible for inclusion

Exclusion Criteria:

* Patient refusal
* Contraindication to nasal swabbing (arm 1)
* Allergy/sensitivity to chlorhexidine gluconate (CHG) (arm 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1518 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marci Drees, MD, MS, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Hospital, Newark, Delaware, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Surveillance Cultures: Active surveillance cultures (via nasal swabs) will be performed for all patients admitted to the medical ICU during the designated study period. Participants will remain in contact isolation until results return as negative.
- Chlorhexidine Gluconate (CHG): Chlorhexidine gluconate (CHG) cloths will be used to bathe patients daily instead of standard soap and water. Active surveillance cultures will also be performed but results will be blinded for duration of study and will not be used to determine need for contact isolation.
Period: Overall Study
Arm/Group | Active Surveillance Cultures | Chlorhexidine Gluconate (CHG)
Started | 750 | 768
Completed | 717 | 715
Not Completed | 33 | 53
Not completed — Missing sufficient data for analysis | 33 | 53

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Surveillance Cultures | Chlorhexidine Gluconate (CHG) | Total
Number analyzed (Participants) | 750 | 768 | 1518
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 405 | 438 | 843
  >=65 years | 345 | 330 | 675
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (15) | 60 (15) | 61 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 390 | 384 | 774
  Male | 360 | 384 | 744
Region of Enrollment [Number; unit: participants]
  United States | 750 | 768 | 1518

OUTCOME MEASURES:

1. Primary Outcome: Acquisition of Methicillin-resistant Staph Aureus (MRSA) Colonization or Infection
Description: Number of patients who acquired MRSA by the time of ICU discharge (based on nasal swab or clinical culture).
Time Frame: During ICU stay
Population: For this observational study, subjects were considered at risk for MRSA acquisition if they had no prior history of MRSA, did not have an MRSA infection that was present on admission, and had an ICU length of stay of at least 48 hours.
Measure: Number; unit: participants
Groups:
- Active Surveillance Cultures (ASC): Active surveillance cultures (via nasal swabs) will be performed for all patients admitted to the medical ICU during the designated study period. Patient will remain in contact isolation until results returned as negative.
- Chlorhexidine Gluconate (CHG): Chlorhexidine gluconate (CHG) cloths will be used to bathe patients daily instead of standard soap and water. Active surveillance cultures will be performed but results will be blinded and not used to determine need for contact isolation.
Arm/Group | Active Surveillance Cultures (ASC) | Chlorhexidine Gluconate (CHG)
Number analyzed (Participants) | 347 | 340
participants | 9 | 10
Statistical Analysis 1: Comparison: Active Surveillance Cultures (ASC) vs Chlorhexidine Gluconate (CHG); Null hypothesis was that ASC and CHG would be no different in preventing acquisition of MRSA; Test type: Superiority or Other; p > 0.05, Regression, Logistic; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.5 to 2.9]

2. Secondary Outcome: Number of Participants With Central Line Associated Bloodstream Infection
Time Frame: During ICU stay up to six months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Active Surveillance Cultures (ASC) | Chlorhexidine Gluconate (CHG)
Number analyzed (Participants) | 347 | 340
participants | 5 | 3

3. Secondary Outcome: Vancomycin Resistant Enterococcal Infection or Colonization
Time Frame: During ICU stay
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance Cultures (ASC) | Chlorhexidine Gluconate (CHG)
Number analyzed (Participants) | 347 | 340
Participants | 7 | 4

ADVERSE EVENTS:
Arm/Group | Active Surveillance Cultures | Chlorhexidine Gluconate (CHG)
Serious Adverse Events (participants affected / at risk) | 0/750 | 0/768
Other Adverse Events (participants affected / at risk) | 0/750 | 0/768

LIMITATIONS AND CAVEATS:
* Single-center, single-unit study limits generalizability
* MRSA acquisition rates lower during both intervention groups than expected, resulting in under-powering of study
* Baseline rate of acquisition of colonization unknown

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No